CLINICAL TRIAL: NCT02559232
Title: An Observational Cross-sectional Study Evaluating the Use of Re-sources and the Sociodemographic and Clinical Characteristics of Patients Diagnosed With NVAF With a Risk of Stroke or Systemic Embolism on Anticoagulant Therapy and Treated in Primary Care Centers
Brief Title: An Observational Cross-sectional Study Evaluating the Use of Re-sources and the Sociodemographic and Clinical Characteristics of Patients Diagnosed With Non-valvular Atrial Fibrillation With a Risk of Stroke or Systemic Embolism on Anticoagulant Therapy and Treated in Primary Care Centers
Acronym: BRONCE-AP
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17961
Record Dates: First submitted 2015-09-17; First posted 2015-09-24 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Stroke; Prevention and Control; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DOAC treated patients: Patients diagnosed with Non-Valvular Atrial Fibrillation at risk of stroke or systemic embolism treated in primary care centres with DOAC.
  Interventions: Drug: Direct Oral Anticoagulant (DOAC)

INTERVENTIONS:
Drug: Direct Oral Anticoagulant (DOAC) — Treatment pattern following the summary of product characteristics

SUMMARY:
This is a retrospective observational study to describe the sociodemographic and clinical characteristics of patients diagnosed with non-valvular atrial fibrillation (NVAF) at risk of stroke or systemic embolism, who at least three months ago changed their anticoagulant therapy, due to any clinical situation, and are currently on treatment with a direct oral anticoagulant (DOAC)

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age diagnosed with non-valvular atrial fibrillation with a risk of stroke or systemic embolism treated in primary care centres.
* Patients on regular treatment with anticoagulants who have changed their therapeutic regimen due to any clinical situation and have been on treatment with a direct oral anticoagulant for at least three months before being recruited (date of signing the in-formed consent).
* Patients whose first direct oral anticoagulant prescription is written by the specialist (cardiologist, haematologist, internist, etc.) and who are followed in primary care.
* Patients who have given their informed consent in writing.

Exclusion Criteria:

* Patients who changed their anticoagulant therapy within a period of less than three months before signing the informed consent.
* Patients with cognitive impairment preventing them from understanding what is written in the patient information sheet or the informed consent, or from per-forming the self-administered questionnaires.
* Patients who started anticoagulant therapy for non-valvular atrial fibrillation with a direct oral anticoagulant .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at risk of stroke or systemic embolism on anticoagulant therapy, who have changed their therapeutic regimen according to their doctor's decision, due to any clinical situation and based on routine clinical practice, and who at the time of enrolment in the study have been receiving treatment with a DOAC for at least three months
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Age | At baseline visit
  sociodemographic data
Gender | At baseline visit
  sociodemographic data
Race | At baseline visit
  sociodemographic data
Composite of relevant cardiovascular events: stroke, TIA, systemic embolism, bleeding | At baseline visit
  sociodemographic data
Composite number of participants with comorbidities: hypertension, heart failure, diabetes mellitus, kidney failure, dyslipidemia | At baseline visit
  clinical characteristics
Dose on the Non-Valvular Atrial Fibrillation treatment: relevant active substances | At baseline visit
  clinical characteristics
Frequency on the Non-Valvular Atrial Fibrillation treatment: relevant active substances | At baseline visit
  clinical characteristics
Duration on the Non-Valvular Atrial Fibrillation treatment: relevant active substances | At baseline visit
  clinical characteristics
Concomitant treatments: therapy group of relevant active substances | At baseline visit
  clinical characteristics; therapy group of relevant active substances: antiarrhythmics, Angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers, β-blockers, dihydropyridine calcium channel blockers, diuretics, hypolipemiant drugs, oral anti-diabetics and human insulin, antiplatelet agents, nonsteroidal anti-inflammatory drugs, Proton-pump inhibitors, others: specify
Risk of thromboembolic event based on the CHADS2 score | At baseline visit
  clinical characteristics; CHADS2: Cardiac failure, Hypertension, Age, Diabetes, Stroke
Risk of thromboembolic event based on the CHA2DS2-VASc score | At baseline visit
  clinical characteristics; CHA2DS2-VASc:Cardiac failure, Hypertension, Age ≥75, Diabetes, Stroke -Vascular disease, Age and sex category
Risk of bleeding based on the HAS-BLED score | At baseline visit
  clinical characteristics; HAS-BLED: Hypertension, Abnormal renal/liver function, Stroke, Bleeding history or predisposition, Labile INR, Elderly , Drugs/alcohol concomitantly

SECONDARY OUTCOMES:
Adherence to treatment | At baseline visit
  use of Haynes-Sackett test
Satisfaction of treatment by the mean score on the ACTS (Anti Clot Treatment Scale) questionnaire | At baseline visit
Compliance with the criteria in therapeutic positioning report UT/V4/23122013 | At baseline visit
  In some Spanish regions it is mandatory to accomplish the conditions of the national guideline UT/V4/23122013 regarding the use of direct oral anticoagulant. In that guideline the characteristics of patients candidates to direct oral anticoagulant are explained.
Use of healthcare resources: Number of visits with primary care physician. Number of visits with specialist, Number of visits with nursing staff, Number of visits to A&E, Number of diagnostic tests in the period when the change was made, related to NVAF. | At baseline visit
  Healthcare resources

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Spain